CLINICAL TRIAL: NCT01144585
Title: Effects of Remote Ischemic Preconditioning and Postconditioning on Lung Ischemic-reperfusion Injury During Cardiopulmonary Bypass - Substudy of NCT00997217
Brief Title: Effects of Remote Ischemic Preconditioning and Postconditioning on Lung Injury During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-1001-016-306
Record Dates: First submitted 2010-06-09; First posted 2010-06-15 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Acute Lung Injury
Keywords: RIPC; lung protection; ischemic reperfusion injury; cardiopulmonary bypass
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC (Experimental): those who receive RIPC and RIPoC before and after CPB
  Interventions: Procedure: remote ischemic preconditioning and postconditioning
- Control (Placebo Comparator): this group have same pneumatic cuff around their arm, but it is not inflated.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: remote ischemic preconditioning and postconditioning — RIPC is done before the use of CPB. It consists of 4 cycles of 5 minutes inflation of pneumatic cuff to 200 mmHg and deflation for 5 minutes. RIPoC is exactly same procedure done "after" CPB.
  Arms: RIPC
Procedure: Control — This group has same pneumatic cuff during the surgery, but it is not inflated during the surgery
  Arms: Control

SUMMARY:
Remote Ischemic Preconditioning(RIPC) and remote ischemic postconditioning(RIPoC) seems to have a protective effect during ischemic period. Using cardiopulmonary bypass(CPB) during open heart surgery reduces pulmonary blood flow and may cause ischemic damage to lung tissue. The investigators anticipate that RIPC and RIPoC may reduce lung injury after CPB.

DETAILED DESCRIPTION:
Cardiopulmonary bypass(CPB) can cause lung function deterioration through various mechanisms. Lung parenchymal tissue ischemia resulted by pulmonary atelectasis and decreased bronchial circulation during CPB is one of the reasons. There were few studies reported that RIPC and RIPoCcan benefit lung function of children or infant after CPB, but studies about adults are still lacking.

Purpose:

The purpose of this study is to evaluate effect of RIPC and RIPoC on the lung function after CPB.

Methods:

Patients will randomly allocated either in study group or control group. Study group will receive RIPC and RIPoC maneuver before and after CPB. Control group will have same automated cuff around their arm but it will not activated. Care givers will be blinded whether the automated cuff is on or not.

We will compare pulmonary parameters (PaO2/FiO2, dynamic and static compliances, Intrapulmonary shunts, etc.) between study group and control group, and check levels of plasma cytokines(IL-4, IL-8, IL-10, TNF-alpha) till 24hr after the operation.

ELIGIBILITY:
Inclusion Criteria:

* those who aged 18-80 years old and planned to undergo elective open heart surgery using cardiopulmonary bypass

Exclusion Criteria:

* emergent operation
* preoperative use of inotropics or mechanical assist device,
* left ventricular ejection fraction less than 30%,
* severe liver, renal disease,
* recent myocardial infarction (within 7 days),
* recent systemic infection or sepsis (within 7 days)
* peripheral vascular disease affecting upper limbs
* amputation of the upper limbs
* major combined operation such as aortic surgery or carotid endarterectomy
* descending thoracic aortic surgery
* rare surgeries; cardiac transplantation, correction of complicated congenital anomalies, pulmonary thromboembolectomy, etc
* significantly decreased pulmonary function before the planned surgery (e.g. using ventilator, oxygen therapy, tachypnea, orthopnea, active lung lesion on chest X-ray, FEV1/FVC less than 50% of predicted level, PaO2 less than 80 mmHg)
* intracardiac shunt
* severe pulmonary artery hypertension
* systemic or local steroid therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
arterial partial pressure of oxygen divided by fraction of inspired oxygen | within 24hr after the surgery
  follow up PaO2/FiO2 during operation and after the opreation for 24 hours

SECONDARY OUTCOMES:
plasma cytokines | within 24hr after the surgery
  follow up plasma IL-6, IL-8, IL-10, TNF-alpha levels during the surgery and within 24hr after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: YunSeok Jeon, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea